CLINICAL TRIAL: NCT02545725
Title: Quality of Life in (ex-)Cancer Patients, Based on the Belgian Cancer Registry. Pilot Study: Quality of Life in Colorectal (ex-)Cancer Patients.
Brief Title: Quality of Life in Colorectal (ex-)Cancer Patients, Based on the Belgian Cancer Registry.
Acronym: QOLColorect
Status: Completed | Type: Observational
Sponsor: Elizabeth Van Eycken (Other)
Collaborators: Flemish League Against Cancer (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Van Eycken, Director Belgian Cancer Registry, Belgian Cancer Registry
Organization: Belgian Cancer Registry (Other)
Other Study IDs: S57073
Record Dates: First submitted 2015-09-01; First posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer; Quality of Life
Keywords: Colorectal Cancer; Quality of life; Questionnaires
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaire on Quality of Life — The patients were asked to complete a questionnaire on Quality of Life

SUMMARY:
This study is collecting data on quality of life, (care)needs and socio-economic factors in colorectal (ex-)cancer patients via a written questionnaire completed by the patient him/herself. The collected data will be linked with the patient- and tumour characteristics available in the database of the Belgian Cancer Registry and with the facturation data supplying information about diagnostic techniques and performed treatments (available via the insurance companies).

Based on the selection criteria, 1220 patients were finally selected from the database of the Belgian Cancer Registry. These patients received an invitation letter by regular mail, a detailed questionnaire and an informed consent.

The questionnaire contains topics as sociodemographic, life style, comorbidity, satisfaction with the provided information, care needs, quality of life, anxiety and depression, financial situation etc.

The patients were asked to complete the questionnaire and send it back, together with the signed informed consent, to the study-collaborators.

After 2-4 weeks, a reminder was sent. At that time, a reply card was added. If a patient doesn't want to participate in this study, a reason can be mentioned on the reply card.

The collected data are linked with the clinical data. The dataset will be coded before analyses will start.

ELIGIBILITY:
Inclusion Criteria:

* Invasive colorectal cancer (ICD-10: C18-C19-C20)
* Patient knows his/her diagnosis of cancer
* Incidence in 2008, 2009 or 2010
* The patient is at least 18 years at diagnosis
* The patient is maximal 90 years when completing the questionnaire
* The patient lives in Flanders and speaks Dutch
* The patient is treated/followed by 1 of the 7 participating hospitals
* The patient is able to complete the questionnaire him/herself (no cognitive problems)

Exclusion Criteria:

* More than 1 invasive tumour diagnosed

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of colorectal cancer (ICD-10: C18-C19-C20) with incidence in 2008-2010 were selected for this study. Patients are at least 18 years old at diagnosis and maximal 90 years old when completing the questionnaire.
  Patients are living in Flanders, speak Dutch and are followed in 1 of the 7 participating hospitals.
  The patients are able to complete the questionnaire themselves: patients with cognitive problems are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1220 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Questionnaire on Quality of Life | 5-8 years after diagnosis
Questionnaire on Quality of Life | At the moment of diagnosis and primary treatment (until +/- 1 year after diagnosis)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Van Eycken, Study Director — Director Belgian Cancer Registry
Locations (1):
- Belgian Cancer Registry, Brussels, Koningsstraat 215 B7, Belgium

REFERENCES:
- See also: Belgian Cancer Registry — http://www.kankerregister.org